CLINICAL TRIAL: NCT04876937
Title: Low-Dose Dexmedetomidine for Delirium Prevention in Mechanically Ventilated Septic Patients in Intensive Care Unit: a Multi-Center, Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: Low-Dose Dexmedetomidine for Delirium Prevention in Mechanically Ventilated Septic Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The trial was stopped prematurely because of slow recruitment.
Sponsor: Peking University First Hospital (Other)
Collaborators: China-Japan Friendship Hospital (Other); Beijing Hospital (Other Government); Beijing Friendship Hospital (Other); Beijing Shijitan Hospital, Capital Medical University (Other); Beijing Tongren Hospital (Other)
Responsible Party: Principal Investigator, Dong-Xin Wang, Professor and Chairman, Department of Anesthesiology and Critical Care Medicine, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2020-241
Record Dates: First submitted 2021-05-03; First posted 2021-05-07 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Adult; Intensive Care Unit; Sepsis; Mechanical Ventilation; Delirium; Dexmedetomidine
Keywords: Adult; Intensive care unit; Sepsis; Mechanical ventilation; Delirium; Dexmedetomidine
MeSH Terms: conditions — Sepsis; Delirium | interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine group (Experimental): Dexmedetomidine is infused at a rate of 0.1-0.2 ug/kg/h during mechanical ventilation, for a maximum of 7 days.
  Interventions: Drug: Dexmedetomidine
- Placebo group (Placebo Comparator): Placebo (normal saline) is infused at a same rate as in the dexmedetomidine group during mechanical ventilation, for a maximum of 7 days.
  Interventions: Drug: Placebo (normal saline)

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine is infused at a rate of 0.1-0.2 μg/kg/h (0.025-0.05 ml/kg/h) from study recruitment in the ICU during mechanical ventilation, for no more than 7 days.
  Other Names: Dexmedetomidine hydrochloride
  Arms: Dexmedetomidine group
Drug: Placebo (normal saline) — Placebo (normal saline) is infused at a rate of 0.025-0.05 ml/kg/h from study recruitment in the ICU during mechanical ventilation, for no more than 7 days.
  Other Names: Normal saline
  Arms: Placebo group

SUMMARY:
Delirium is common in septic patients, especially those receiving mechanical ventilation in the intensive care unit (ICU). Dexmedetomidine is a highly selective α2 adrenoreceptor agonist with anxiolytic, sedative, analgesic, and anti-inflammatory effects. Use of dexmedetomidine in mechanically ventilated ICU patients is associated with less delirium and improved outcomes. However, dexmedetomidine infusion produces dose-dependent bradycardia and hypotension; these limited the use of dexmedetomidine in ICU patients. This study is designed to test the hypothesis that low-dose dexmedetomidine infusion can also reduce delirium in mechanically ventilated ICU patients with sepsis.

DETAILED DESCRIPTION:
Delirium is an acutely occurred and fluctuating disorder of consciousness, attention, and cognition. The occurrence of delirium is associated with worse outcomes including prolonged mechanical ventilation, prolonged length of stay in ICU and hospital, increased complications, higher in-hospital mortality, and evaluated medical expenses. It is also associated with worse long-term outcomes including cognitive decline, worse quality of life, and shortened long-term survival.

Dexmedetomidine is a highly selective α2 adrenoreceptor agonist with anxiolytic, sedative, analgesic, and anti-inflammatory effects. Studies showed that use of dexmedetomidine is associated with less delirium in ICU patients. Potential mechanisms may include better sleep quality, less consumption of opioids and benzodiazepines, and suppressed inflammatory response.

The incidence of sepsis in ICU patients is as high as 47.2%; 93% of septic patients relying on mechanical ventilation. Delirium is common in septic patients; the reported incidences varies from 20% to 50%. The incidence of delirium in critically ill patients with mechanical ventilation is up to 60-84%. However, the majority of mechanically ventilated ICU patients are sedated with propofol; only 10% of them are given dexmedetomidine. A main reason is that dexmedetomidine infusion is associated with dose-related bradycardia and hypotension.

In a previous study, might-time low-dose dexmedetomidine infusion (0.1 μg/kg/h) improved subjective sleep quality and reduced delirium in elderly patients admitted to ICU after surgery. In another study of ICU patients receiving mechanical ventilation, low-dose dexmedetomidine infusion (0-0.5 μg/kg/h) based on protocol sedation also reduced delirium and shortened mechanical ventilation without increasing adverse events. We hypothesized that, in ICU septic patients with mechanical ventilation, low-dose dexmedetomidine infusion (0.1-0.2 μg/kg/h) might also reduce delirium.

The purpose of this study is to investigate the effect of low-dose dexmedetomidine infusion on incidence of delirium in ICU septic patients with mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older;
2. Admitted to the ICU;
3. With expected mechanical ventilation duration ≥12 hours;
4. Meet the diagnostic criteria of sepsis (sepsis 3.0; patient with infection and a sequential organ failure assessment score ≥2).

Exclusion Criteria:

1. Refuse to participate in;
2. Pregnancy;
3. History of schizophrenia, epilepsy, parkinsonism, or myasthenia gravis;
4. Inability to communicate (coma, profound dementia, or language barrier);
5. Brain injury or neurosurgery;
6. Left ventricular ejection fraction (LVEF) less than 30%, sick sinus syndrome, severe sinus bradycardia (<50 beats per min [bpm]), or second degree or greater atrioventricular block without pacemaker;
7. Serious hepatic dysfunction (Child-Pugh class C);
8. Serious renal dysfunction (undergoing dialysis);
9. With expected survival for no more than 24 hours;
10. Allergic to dexmedetomidine;
11. Other conditions that were considered unsuitable for study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-05-28 (Actual); Primary Completion 2024-02-02 (Actual); Study Completion 2024-03-02 (Actual)

PRIMARY OUTCOMES:
Incidence of delirium within the first 7 days after enrollment | Up to 7 days after enrollment
  Delirium is assessed twice daily (from 06:00 to 10:00 and from 18:00 to 20:00) with the Confusion Assessment Method for the intensive care unit (CAM-ICU).

SECONDARY OUTCOMES:
Duration of mechanical ventilation. | Up to 30 days after enrollment
  Duration of mechanical ventilation after study enrollment.
Length of stay in the ICU. | Up to 30 days after enrollment
  Length of stay in the ICU after study enrollment.
Length of stay in the hospital. | Up to 30 days after enrollment
  Length of stay in the hospital after study enrollment.
Incidence of non-delirium complications. | Up to 30 days after enrollment
  Non-delirium complications are defined as newly occurred medical conditions other than delirium that required therapeutic intervention, i.e., grade 2 or higher on Clavien-Dindo classification.
All-cause 30-day mortality | Up to 30 days after enrollment
  All-cause 30-day mortality after study enrollment.
30-day cognitive function | On the 30th day after enrollment.
  Cognitive function is assessed with the Modified Telephone Interview for Cognitive Status (TICS-m) which is a 12-item questionnaire that verbally assesses global cognitive function via telephone. The score ranges from 0 to 50, with higher score indicating better function.
30-day quality of life | On the 30th day after enrollment.
  Quality-of-life is assessed with the World Health Organization Quality of Life brief version (WHOQOL-BREF) which is a 24-item questionnaire that assesses the quality of life in physical, psychological, and social relationship, and environmental domains. The score ranges from 0 to 100 for each domain, with higher score indicating better function.

OTHER OUTCOMES:
Pain intensity. | Up to 7 days after enrollment.
  Assessed twice daily (from 06:00 to 10:00 and from 18:00 to 20:00) with the Numeric Rating Scale (NRS, an 11-point scale where 0 indicated no pain and 10 indicated the worst possible pain).
Subjective sleep quality. | Up to 7 days after enrollment.
  Assessment once daily (from 06:00 to 10:00) with the Numeric Rating Scale (NRS, an 11-point scale where 0 indicated the best possible sleep and 10 indicated the worst possible sleep).
Score of Acute Physiology and Chronic Health Evaluation II (APACHE II). | Within 24 hours after enrollment.
  Score of Acute Physiology and Chronic Health Evaluation II (APACHE II).
6-month cognitive function. | At the end of 6 months after enrollment.
  Cognitive function is assessed with the Modified Telephone Interview for Cognitive Status (TICS-m) which is a 12-item questionnaire that verbally assesses global cognitive function via telephone. The score ranges from 0 to 50, with higher score indicating better function.
6-month quality of life. | At the end of 6 months after enrollment.
  Quality-of-life is assessed with the World Health Organization Quality of Life brief version (WHOQOL-BREF) which is a 24-item questionnaire that assesses the quality of life in physical, psychological, and social relationship, and environmental domains. The score ranges from 0 to 100 for each domain, with higher score indicating better function.
Overall survival | Up to 1 year after enrollment.
  Overall survival
1-year cognitive function. | At the end of 1 year after enrollment.
  Cognitive function is assessed with the Modified Telephone Interview for Cognitive Status (TICS-m) which is a 12-item questionnaire that verbally assesses global cognitive function via telephone. The score ranges from 0 to 50, with higher score indicating better function.
1-year quality of life. | At the end of 1 year after enrollment.
  Quality-of-life is assessed with the World Health Organization Quality of Life brief version (WHOQOL-BREF) which is a 24-item questionnaire that assesses the quality of life in physical, psychological, and social relationship, and environmental domains. The score ranges from 0 to 100 for each domain, with higher score indicating better function.

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, MD,PhD, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guenther U, Radtke FM. Delirium in the postanaesthesia period. Curr Opin Anaesthesiol. 2011 Dec;24(6):670-5. doi: 10.1097/ACO.0b013e32834c7b44. PMID 21971396
- [Background] Roberts B, Rickard CM, Rajbhandari D, Turner G, Clarke J, Hill D, Tauschke C, Chaboyer W, Parsons R. Multicentre study of delirium in ICU patients using a simple screening tool. Aust Crit Care. 2005 Feb;18(1):6, 8-9, 11-4 passim. doi: 10.1016/s1036-7314(05)80019-0. PMID 18038529
- [Background] Ely EW, Gautam S, Margolin R, Francis J, May L, Speroff T, Truman B, Dittus R, Bernard R, Inouye SK. The impact of delirium in the intensive care unit on hospital length of stay. Intensive Care Med. 2001 Dec;27(12):1892-900. doi: 10.1007/s00134-001-1132-2. Epub 2001 Nov 8. PMID 11797025
- [Background] Balas MC, Happ MB, Yang W, Chelluri L, Richmond T. Outcomes Associated With Delirium in Older Patients in Surgical ICUs. Chest. 2009 Jan;135(1):18-25. doi: 10.1378/chest.08-1456. Epub 2008 Nov 18. PMID 19017895
- [Background] Ansaloni L, Catena F, Chattat R, Fortuna D, Franceschi C, Mascitti P, Melotti RM. Risk factors and incidence of postoperative delirium in elderly patients after elective and emergency surgery. Br J Surg. 2010 Feb;97(2):273-80. doi: 10.1002/bjs.6843. PMID 20069607
- [Background] Ely EW, Shintani A, Truman B, Speroff T, Gordon SM, Harrell FE Jr, Inouye SK, Bernard GR, Dittus RS. Delirium as a predictor of mortality in mechanically ventilated patients in the intensive care unit. JAMA. 2004 Apr 14;291(14):1753-62. doi: 10.1001/jama.291.14.1753. PMID 15082703
- [Background] Franco K, Litaker D, Locala J, Bronson D. The cost of delirium in the surgical patient. Psychosomatics. 2001 Jan-Feb;42(1):68-73. doi: 10.1176/appi.psy.42.1.68. PMID 11161124
- [Background] Abelha FJ, Luis C, Veiga D, Parente D, Fernandes V, Santos P, Botelho M, Santos A, Santos C. Outcome and quality of life in patients with postoperative delirium during an ICU stay following major surgery. Crit Care. 2013 Oct 29;17(5):R257. doi: 10.1186/cc13084. PMID 24168808
- [Background] Van Rompaey B, Schuurmans MJ, Shortridge-Baggett LM, Truijen S, Elseviers M, Bossaert L. Long term outcome after delirium in the intensive care unit. J Clin Nurs. 2009 Dec;18(23):3349-57. doi: 10.1111/j.1365-2702.2009.02933.x. Epub 2009 Sep 4. PMID 19735334
- [Background] Bickel H, Gradinger R, Kochs E, Forstl H. High risk of cognitive and functional decline after postoperative delirium. A three-year prospective study. Dement Geriatr Cogn Disord. 2008;26(1):26-31. doi: 10.1159/000140804. Epub 2008 Jun 24. PMID 18577850
- [Background] Pisani MA, Kong SY, Kasl SV, Murphy TE, Araujo KL, Van Ness PH. Days of delirium are associated with 1-year mortality in an older intensive care unit population. Am J Respir Crit Care Med. 2009 Dec 1;180(11):1092-7. doi: 10.1164/rccm.200904-0537OC. Epub 2009 Sep 10. PMID 19745202
- [Background] Kawazoe Y, Miyamoto K, Morimoto T, Yamamoto T, Fuke A, Hashimoto A, Koami H, Beppu S, Katayama Y, Itoh M, Ohta Y, Yamamura H; Dexmedetomidine for Sepsis in Intensive Care Unit Randomized Evaluation (DESIRE) Trial Investigators. Effect of Dexmedetomidine on Mortality and Ventilator-Free Days in Patients Requiring Mechanical Ventilation With Sepsis: A Randomized Clinical Trial. JAMA. 2017 Apr 4;317(13):1321-1328. doi: 10.1001/jama.2017.2088. PMID 28322414
- [Background] Wunsch H, Kahn JM, Kramer AA, Wagener G, Li G, Sladen RN, Rubenfeld GD. Dexmedetomidine in the care of critically ill patients from 2001 to 2007: an observational cohort study. Anesthesiology. 2010 Aug;113(2):386-94. doi: 10.1097/ALN.0b013e3181e74116. PMID 20613466
- [Background] van Vught LA, Klein Klouwenberg PM, Spitoni C, Scicluna BP, Wiewel MA, Horn J, Schultz MJ, Nurnberg P, Bonten MJ, Cremer OL, van der Poll T; MARS Consortium. Incidence, Risk Factors, and Attributable Mortality of Secondary Infections in the Intensive Care Unit After Admission for Sepsis. JAMA. 2016 Apr 12;315(14):1469-79. doi: 10.1001/jama.2016.2691. PMID 26975785
- [Background] Nelson LE, Lu J, Guo T, Saper CB, Franks NP, Maze M. The alpha2-adrenoceptor agonist dexmedetomidine converges on an endogenous sleep-promoting pathway to exert its sedative effects. Anesthesiology. 2003 Feb;98(2):428-36. doi: 10.1097/00000542-200302000-00024. PMID 12552203
- [Background] Djaiani G, Silverton N, Fedorko L, Carroll J, Styra R, Rao V, Katznelson R. Dexmedetomidine versus Propofol Sedation Reduces Delirium after Cardiac Surgery: A Randomized Controlled Trial. Anesthesiology. 2016 Feb;124(2):362-8. doi: 10.1097/ALN.0000000000000951. PMID 26575144
- [Background] Su X, Meng ZT, Wu XH, Cui F, Li HL, Wang DX, Zhu X, Zhu SN, Maze M, Ma D. Dexmedetomidine for prevention of delirium in elderly patients after non-cardiac surgery: a randomised, double-blind, placebo-controlled trial. Lancet. 2016 Oct 15;388(10054):1893-1902. doi: 10.1016/S0140-6736(16)30580-3. Epub 2016 Aug 16. PMID 27542303
- [Background] Reade MC, Eastwood GM, Bellomo R, Bailey M, Bersten A, Cheung B, Davies A, Delaney A, Ghosh A, van Haren F, Harley N, Knight D, McGuiness S, Mulder J, O'Donoghue S, Simpson N, Young P; DahLIA Investigators; Australian and New Zealand Intensive Care Society Clinical Trials Group. Effect of Dexmedetomidine Added to Standard Care on Ventilator-Free Time in Patients With Agitated Delirium: A Randomized Clinical Trial. JAMA. 2016 Apr 12;315(14):1460-8. doi: 10.1001/jama.2016.2707. PMID 26975647
- [Background] Geloen A, Chapelier K, Cividjian A, Dantony E, Rabilloud M, May CN, Quintin L. Clonidine and dexmedetomidine increase the pressor response to norepinephrine in experimental sepsis: a pilot study. Crit Care Med. 2013 Dec;41(12):e431-8. doi: 10.1097/CCM.0b013e3182986248. PMID 23963131
- [Background] Brummel NE, Jackson JC, Pandharipande PP, Thompson JL, Shintani AK, Dittus RS, Gill TM, Bernard GR, Ely EW, Girard TD. Delirium in the ICU and subsequent long-term disability among survivors of mechanical ventilation. Crit Care Med. 2014 Feb;42(2):369-77. doi: 10.1097/CCM.0b013e3182a645bd. PMID 24158172